CLINICAL TRIAL: NCT04505787
Title: Characterisation of Relative Bioavailability of a Newly Developed S-flurbiprofen Containing Patch Formulation in Comparison With a Marketed Oral Flurbiprofen Containing Tablet Formulation - a Multiple Dose, Randomised, 2-period Crossover...
Brief Title: S-flurbiprofen Bioavailability Trial to Compare a Newly Developed Patch vs. a Marketed Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SocraTec R&D GmbH (Other)
Collaborators: Teikoku Seiyaku Co., Ltd. (Industry); SocraMetrics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1378fbp19ct; 2019-003918-14 (EudraCT Number); TK-254R-0101 (Other: Client protocol number (Teikoku Seiyaku Co.))
Record Dates: First submitted 2020-07-13; First posted 2020-08-10 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Comparative Bioavailability
Keywords: Bioavailability
MeSH Terms: interventions — Flurbiprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Esflurbiprofen hydrogel patch (Experimental): "Esflurbiprofen hydrogel patch 165 mg" (EFHP) (Teikoku Seiyaku Co.), transdermal patch containing 165 mg S-flurbiprofen, once daily consecutive application over 14 days; each patch to be applied for 24 h, application site: outer ankle (same site and position for all applied patches)
  Interventions: Drug: Esflurbiprofen hydrogel patch 165 mg (EFHP)
- Froben (Active Comparator): "Froben 100 mg comprimidos revestidos" (Abbott Laboratórios, Lda., Portugal), immediate release tablets containing 100 mg flurbiprofen, oral multiple dose administration of 1 tablet three times daily (TID) over 4 consecutive days after a light meal
  Interventions: Drug: Froben 100 mg comprimidos revestidos

INTERVENTIONS:
Drug: Esflurbiprofen hydrogel patch 165 mg (EFHP) — patch application with PK blood sampling
  Arms: Esflurbiprofen hydrogel patch
Drug: Froben 100 mg comprimidos revestidos — tablet administration with PK blood sampling
  Arms: Froben

SUMMARY:
Teikoku Seiyaku Co., Ltd. (Japan) is developing a new Esflurbiprofen Hydrogel Patch (EFHP), a transdermal product containing 165 mg of the S-enantiomer of flurbiprofen (S-flurbiprofen) as its active pharmaceutical ingredient.

The present clinical trial will be conducted to characterise maximum observed systemic exposure of the newly developed EFHP (Test) vs. "Froben 100 mg" (Reference, containing 100 mg racemic flurbiprofen in a 1:1 ratio). Characterisation will be performed under steady state conditions in order to bridge the available safety information on the basis of the comparison of maximum observed systemic exposure by means of AUC0-24h,ss,P vs. AUC0-24,ss,T and Cmax,ss,P vs. Cmax,ss,T of S-flurbiprofen.

DETAILED DESCRIPTION:
This single centre, open-label, randomised (order of treatments), balanced, multiple dose trial will be performed in a 2-period, 2-sequence-crossover design.

The Test Product (patch) will be applied once daily over 14 consecutive days, whereby each patch will remain applied for 24 h. Blood sampling will be performed after the 1st patch application over 24 h in order to characterise the single dose application and after the 14th patch application over 72 h in order to characterise pharmacokinetic parameters after multiple dosing including elimination phase. In between through values will be taken in the morning of specified study days to characterise steady-state built-up phase.

The Reference product will be administered after a light meal as single oral doses of 100 mg flurbiprofen three times daily (i.e. every 8 h) over 4 days. Blood sampling will be performed after the 10th tablet administration over 72 h in order to characterise pharmacokinetic parameters after multiple dosing including elimination phase. In between through values will be taken in the morning of study days 1 to 4 to characterise steady-state built-up phase.

The clinical trial will be performed as a cross-over investigation with intra-individual comparison, thus reducing variability of the pharmacokinetic parameters, which is supposed to be higher between subjects than within an individual subject.

ELIGIBILITY:
Inclusion Criteria:

1. age: 18 to 64 years (inclusive)
2. body-mass index (BMI): >= 18.5 kg/m² and <= 30.0 kg/m²
3. good state of health
4. non-smoker or ex-smoker for at least 3 months
5. written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

Safety concerns

1. existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
2. existing or history of hypertension and/or heart failure
3. existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient
4. existing gastrointestinal diseases or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
5. history of gastrointestinal bleeding or perforation related to previous NSAID therapy
6. active, or history of, ulcerative colitis, Crohn's disease, peptic ulceration or gastrointestinal haemorrhage
7. existing metabolic, endocrine and/or immunologic diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient
8. diabetes mellitus
9. hyperlipidaemia (LDL > 160 mg/dL; HDL < 35 mg/dL; triglycerides > 200 mg/dL; cholesterol > 240 mg/dL)
10. history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
11. presence or history of acute or chronic diseases of the skin (e.g. atopy, neurodermatitis, contact allergy, eczema, psoriasis, vitiligo, melanoma, squamous cell carcinoma), any dermatological condition or skin sensitivity which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
12. existing or history of bronchial asthma
13. known allergic reactions (e.g. bronchospasm, rhinitis, angioedema, or urticaria) to the active ingredients used, to acetylsalicylic acid or other NSAIDs, or to constituents of the pharmaceutical preparations
14. history of severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
15. fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency
16. galactose intolerance or Lapp lactase deficiency
17. systolic blood pressure < 90 or > 139 mmHg
18. diastolic blood pressure < 60 or > 89 mmHg
19. heart rate < 50 bpm or > 90 bpm
20. QTc interval > 450 ms for men and > 470 ms for women
21. laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator
22. ASAT > 20% ULN, ALAT > 10% ULN, bilirubin > 20% ULN (except in case of existing Morbus Gilbert-Meulengracht deduced from anamnesis/medical history) and creatinine > 0.1 mg/dL ULN (limit of > 0.1 mg/dL correspondents to of > 9 µmol/l ULN).
23. positive anti-HIV-test (if positive to be verified by western blot), HBs-AG-test or anti-HCV-test
24. symptoms of, or diagnosis of COVID-19 within the last 14 days prior to individual enrolment of the subject
25. contact to persons in risk regions as defined by the Robert Koch Institute within the last 14 days prior to individual enrolment of the subject
26. direct contact to persons with symptoms of, or diagnosis of COVID-19 within the last 14 days prior to individual enrolment of the subject Lack of suitability for the clinical trial
27. skin abnormality (e.g. tattoo (including tattoo that was removed), scar, sunburn or obvious difference in skin colour), open sores, or excessive hair at the application site
28. acute or chronic diseases which may interfere with the pharmacokinetics of the IMP
29. history of or current drug or alcohol dependence
30. positive alcohol or drug test at screening examination
31. regular intake of alcoholic food or beverages of >= 24 g pure ethanol for male or >= 12 g pure ethanol for female per day
32. subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
33. regular intake of caffeine containing food or beverages of >= 500 mg caffeine per day
34. blood donation or other blood loss of more than 400 ml within the last 2 months prior to individual enrolment of the subject
35. administration of any investigational medicinal product during the last 2 months prior to individual enrolment of the subject
36. regular treatment with any systemically available medication (except hormonal contraceptives and hormonal replacement therapy, e.g. estrogens, L-thyroxine)
37. subjects, who report a frequent occurrence of migraine attacks

    For female subjects with childbearing potential only:
38. positive pregnancy test at screening examination
39. pregnant or lactating women
40. female subjects who do not agree to apply highly effective contraceptive methods Administrative reasons
41. subjects suspected or known not to follow instructions
42. subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Assessment of non-superiority of Test in comparison to Reference under steady-state conditions determined by use of AUC0-24,ss,P vs. AUC0-24,ss,T of S-flurbiprofen | 24 hours
  AUC0-24,ss,P = area under the plasma concentration vs. time curve from dosing time to the end of the dosing interval (profiling day after 14th patch application), calculated by means of the linear up/log down method (linear trapezoidal rule for increases in concentration/logarithmic trapezoidal rule for decreases in concentrations AUC0-24,ss,T = area under the plasma concentration vs. time profile over 24 h at profiling day from dosing time of 10th administration to 8 h after 12th administration, calculated by means of the linear up/log down method (linear trapezoidal rule for increases in concentration/logarithmic trapezoidal rule for decreases in concentrations
Assessment of non-superiority of Test in comparison to Reference under steady-state conditions determined by use of Cmax,ss,P vs. Cmax,ss,T of S flurbiprofen | 24 hours
  Cmax,ss,P = maximum concentration in plasma within the dosing interval (profiling day after 14th patch application), obtained directly from measured values Cmax,ss,T = maximum concentration over 24 h at profiling day from dosing time of 10th administration to 8 h after 12th administration, obtained directly from measured values

SECONDARY OUTCOMES:
Skin irritation properties for Esflurbiprofen hydrogel patch by frequency of scores | 16 days
  frequency of scores for local tolerability and skin irritation per time point according to "Assessing the Irritation and Sensitization Potential of Transdermal and Topical Delivery Systems for ANDAs", Guidance for Industry, DRAFT. 2018 October
Patch adhesion properties for Esflurbiprofen hydrogel patch by percentage of adhered patch area | 15 days
  documentation of the percentage of area that remains adhered and scoring (i.e. percentage of adhered area and scores will be matched/combined) per time point according to "Assessing Adhesion With Transdermal and Topical Delivery Systems for ANDAs", Guidance for Industry, DRAFT. 2018 October
Adverse Events | 28 days
  Descriptive characterisation with regard to frequency and intensity, relationship to the IMP, action taken, outcome, and seriousness as well as period and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frank Donath, MD, Principal Investigator — SocraTec R&D GmbH Clinical Pharmacology Unit
Locations (1):
- SocraTec R&D GmbH, Clinical Pharmacology Unit, Erfurt, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: Yes